CLINICAL TRIAL: NCT03824522
Title: Post Marketing Surveillance Study for ADYNOVATE in South Korea
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: Takeda Pharma Korea Co. Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 261603
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BAX 855

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Study Participants: Participants who are newly prescribed with Adynovate and participants previously treated with Adynovate will be treated with ADYNOVATE for hemophilia A at the time of enrollment according to a regimen determined by the study site treating physician.
  Interventions: Biological: ADYNOVATE

INTERVENTIONS:
Biological: ADYNOVATE — Pegylated recombinant human factor VIII
  Other Names: PEGylated rFVIII

SUMMARY:
The main aim of this study is to check for side effects and medical problems in participants with hemophilia A who are receiving ADYNOVATE in routine clinical practice. Also, it will be checked how effective ADYNOVATE is at stopping a bleed, at preventing bleeding episodes when used routinely for prevention and at controlling hemophilia-related bleeding during surgeries.

Participants with hemophilia A who will be newly prescribed with ADYNOVATE treatment or have already been taking ADYNOVATE treatment according to the physician's decision will be included in this study.

Participants will visit the study clinic as a part of their routine clinical practice and will be contacted by phone calls/home visits by home care workers for collection of treatment related data during the 6-month observation period.

ELIGIBILITY:
Inclusion Criteria

Participants with a diagnosis of hemophilia A who will be newly prescribed with ADYNOVATE or already have been prescribed ADYNOVATE according to the study physician's judgment shall be included in this study if:

* The participant or legally authorized representative has given written informed consent to participate in the study.
* The participant is indicated for treatment according to the ADYNOVATE South Korea prescribing information (PI).

Exclusion Criteria

Participants should be excluded from this study if:

* The participant or legally authorized representative does not wish to participate in the study.
* Any of the contraindications included in the PI for ADYNOVATE apply.
* Participant is enrolled in an interventional trial using an investigational product other than ADYNOVATE.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hemophilia A participants in South Korea who will be newly prescribed with ADYNOVATE or already been prescribed with ADYNOVATE will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Throughout the duration of patient participation of up to approximately 6 months
  Serious adverse events and non-serious adverse events
Frequency of adverse events | Throughout the duration of patient participation of up to approximately 6 months
  Serious adverse events and non-serious adverse events

SECONDARY OUTCOMES:
Incidence of inhibitor titers for FVIII antibodies | Throughout the duration of patient participation of up to approximately 6 months
  By titer levels, high and lower titer categories
Number of treated bleeds | Throughout the duration of patient participation of up to approximately 6 months
  Number of treated bleeds throughout the study period
ADYNOVATE units required for bleed resolution | At bleed resolution, throughout the duration of patient participation of up to approximately 6 months
  Number of ADYNOVATE units required for bleed resolution
Number of ADYNOVATE infusions needed for the treatment of bleeding episodes | At bleed resolution, throughout the duration of patient participation of up to approximately 6 months
  The number of ADYNOVATE infusions needed for each bleeding episode is determined by the participant, his/her caregiver, and/or clinician treating the participant, and is based upon the participant's response to treatment
Hemostatic effectiveness assessment of bleeding episodes treated with ADYNOVATE during prophylaxis treatment | Throughout the duration of patient participation of up to approximately 6 months
  Using a 4-point ordinal scale (Excellent, Good, Fair, or None)
Hemostatic effectiveness of ADYNOVATE for participants on an on-demand regimen | At bleed resolution, throughout the duration of patient participation of up to approximately 6 months
  Using a 4-point ordinal scale (Excellent, Good, Fair, or None)
Assessment of perioperative effectiveness of ADYNOVATE | Throughout the duration of patient participation of up to approximately 6 months
  Using a 4-point ordinal scale (Excellent, Good, Fair, or None)
Clinically significant changes in laboratory results | Throughout the duration of patient participation of up to approximately 6 months
  Number of clinically significant changes in laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- South Korea (8):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Severance Hospital Yonsei University Health System, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kim Hugh Chul Internal Medicine, Seoul
  - Korea Hemophilia Foundation (Seoul), Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc74db2bf003ab46012